CLINICAL TRIAL: NCT06772493
Title: ViewFlex X ICE First-in-Human Study
Acronym: ViewFlex X FIH
Status: Recruiting | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: ABT-CIP-10528
Record Dates: First submitted 2025-01-02; First posted 2025-01-13 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Cardiac Arrhythmias
Keywords: Intracardiac Echocardiography; cardiac electrophysiology
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Cohort 1: Single Arm group to undergo a cardiac ablation procedure utilizing the ViewFlex X ICE System
  Interventions: Device: ViewFlex X ICE System
- Cohort 2: Single Arm group to undergo a cardiac ablation procedure utilizing the ViewFlex X ICE System
  Interventions: Device: ViewFlex X ICE System

INTERVENTIONS:
Device: ViewFlex X ICE System — Subjects to undergo cardiac ablation procedure utilizing the ViewFlex X ICE System

SUMMARY:
This prospective, acute, first-in-human, non-significant risk study is intended to evaluate a modified version of the ViewFlex X ICE Catheter, Sensor Enabled (ViewFlex X SE) and ViewMate Multi Ultrasound Console (VMM) ICE data integration with the EnSite X EP System (hereafter referred to as the ViewFlex X ICE System).

ELIGIBILITY:
Inclusion Criteria:

A patient will be eligible for clinical trial participation if they meet the following criteria:

1. Able and willing to provide written informed consent prior to any clinical investigation-related procedure.
2. Plans to undergo any EP procedure utilizing ICE
3. At least 18 years of age

Exclusion Criteria:

A patient will be excluded from enrollment in the study if they meet any of the following criteria:

1. Subject is currently participating in another clinical investigation.
2. Implanted left atrial appendage occluder
3. Implanted mechanical mitral or tricuspid valve replacement
4. Implanted intracardiac device within 30 days
5. Pregnant or nursing
6. Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements, or impact the scientific soundness of the clinical investigation results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This clinical investigation will enroll subjects of all genders over the age of 18 undergoing any previously planned electrophysiology study procedure utilizing ICE.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Physician assessment of the ability to navigate the ViewFlex X SE catheter and adequately visualize major cardiac anatomic structures. | During the procedure
Physician assessment of the ability to use anatomic ICE markers and ICE geometry as a reference during mapping and ablation procedures. | during the procedure
Rate of device- or procedure-related serious adverse events that occur through patient discharge. | during the procedure and periprocedurally

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Ruffner, PhD, Study Director — Abbott
Locations (5):
- United States (5):
  - St. Bernards Medical Center, Jonesboro, Arkansas
  - University of California, San Diego, La Jolla, California
  - Research Medical Center, Kansas City, Missouri
  - NYU Langone Health, New York, New York
  - Medical University of South Carolina, Charleston, South Carolina